CLINICAL TRIAL: NCT02939287
Title: Aprepitant- and Olanzapine- Containing Regimens for Prevention of Acute and Delayed Nausea and Vomiting Associated With High Dose Melphalan and BEAM in Autologous Stem Cell Transplant Patients
Brief Title: Aprepitant- and Olanzapine- Containing Anti-emetic Regimens With High Dose Melphalan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14102001
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Results first posted 2024-01-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Nausea; Vomiting
Keywords: autologous; myeloma; transplant
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms, Plasma Cell | interventions — Aprepitant; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Aprepitant (Active Comparator): aprepitant plus standard anti-emetic regimen
  Interventions: Drug: o Aprepitant 125 mg orally one hour prior to chemotherapy on Day -1 and 80 mg orally on Days 0 and +1
- Olanzapine (Experimental): olanzapine plus standard anti-emetic regimen
  Interventions: Drug: Olanzapine10 mg orally daily on Days -1,0,+1 and +2
- Aprepitant plus olanzapine (Experimental): aprepitant and olanzapine plus standard anti-emetic regimen
  Interventions: Drug: Aprepitant plus Olanzapine

INTERVENTIONS:
Drug: o Aprepitant 125 mg orally one hour prior to chemotherapy on Day -1 and 80 mg orally on Days 0 and +1 — Add aprepitant to anti-emetic regimen
  Other Names: Emend
  Arms: Aprepitant
Drug: Olanzapine10 mg orally daily on Days -1,0,+1 and +2 — add olanzapine to anti-emetic regimen
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Aprepitant plus Olanzapine — add aprepitant and olanzapine to anti-emetic regimen
  Other Names: Emend; Zyprexa
  Arms: Aprepitant plus olanzapine

SUMMARY:
The purpose of this study is to help answer the following research question:

* Whether administration of an aprepitant containing regimen, an olanzapine containing regimen or regimen containing both will prevent nausea and vomiting better for patients undergoing an autologous stem cell transplant with melphalan chemotherapy. Both of these medications are approved by the United States Food and Drug Administration (FDA) for nausea and vomiting.
* Participants will be randomly assigned to one of the 3 treatment groups:

  * Arm A: aprepitant containing anti-emetic therapy
  * Arm B: olanzapine containing anti-emetic therapy
  * Arm C: Aprepitant plus olanzapine containing anti-emetic therapy

DETAILED DESCRIPTION:
This is a multi-center, randomized, non-inferiority phase 3 study conducted to determine an appropriate anti-emetic regimen for patients receiving melphalan for an autologous stem cell transplant (SCT). Candidates for this trial will include patients aged 18-80 years with hematologic malignancies receiving high dose melphalan as part of a conditioning regimen for an autologous stem cell transplant. Patients will be enrolled in 3 arms. Patients in Arm A will receive an aprepitant containing anti-emetic regimen. Patients in Arm B will receive an olanzapine containing anti-emetic regimen. Patients in Arm C will receive an aprepitant plus olanzapine containing anti-emetic regimen. Patients must be able to tolerate oral medications.

Patients will be carefully monitored for rates of emesis, nausea, and mucositis. Any adverse events will be recorded. Impact on quality of life will also be assessed. A total of 184 patients will be accrued to each arm. It is anticipated that the accrual period will last approximately 2-3 years. The primary endpoint of this study is a complete response, defined as no emesis and no rescue therapy within 120 hours of melphalan administration.

ELIGIBILITY:
Inclusion Criteria:

* Autologous transplant containing high dose melphalan as part of the conditioning regimen (single or 2 day melphalan; BEAM [carmustine, etoposide, cytarabine, melphalan])
* able to tolerate oral medications

Exclusion Criteria:

* Nausea/vomiting within 12 hours before planned high dose conditioning chemotherapy
* Any anti-emetic treatment within 24 hours before planned high dose conditioning chemotherapy
* Pregnancy
* Baseline corrected QT interval (QTc) > 500 ms
* History of seizures
* History of central nervous system (CNS) disease
* Human immunodeficiency virus (HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schultz, PharmD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Prestrud AA, Hesketh PJ, Kris MG, Feyer PC, Somerfield MR, Chesney M, Clark-Snow RA, Flaherty AM, Freundlich B, Morrow G, Rao KV, Schwartz RN, Lyman GH; American Society of Clinical Oncology. Antiemetics: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2011 Nov 1;29(31):4189-98. doi: 10.1200/JCO.2010.34.4614. Epub 2011 Sep 26. PMID 21947834
- [Background] Navari RM, Gray SE, Kerr AC. Olanzapine versus aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a randomized phase III trial. J Support Oncol. 2011 Sep-Oct;9(5):188-95. doi: 10.1016/j.suponc.2011.05.002. Epub 2011 Sep 24. PMID 22024310
- [Background] Giralt SA, Mangan KF, Maziarz RT, Bubalo JS, Beveridge R, Hurd DD, Mendoza FL, Rubenstein EB, DeGroot TJ, Schuster MW. Three palonosetron regimens to prevent CINV in myeloma patients receiving multiple-day high-dose melphalan and hematopoietic stem cell transplantation. Ann Oncol. 2011 Apr;22(4):939-946. doi: 10.1093/annonc/mdq457. Epub 2010 Oct 8. PMID 20935058
- [Background] Slaby J, Trneny M, Prochazka B, Klener P. Antiemetic efficacy of three serotonin antagonists during high-dose chemotherapy and autologous stem cell transplantation in malignant lymphoma. Neoplasma. 2000;47(5):319-22. PMID 11130251
- [Background] Ballen KK, Hesketh AM, Heyes C, Becker PS, Emmons RV, Fogarty K, LaPointe J, Liu Q, Hsieh CC, Hesketh PJ. Prospective evaluation of antiemetic outcome following high-dose chemotherapy with hematopoietic stem cell support. Bone Marrow Transplant. 2001 Dec;28(11):1061-6. doi: 10.1038/sj.bmt.1703280. PMID 11781617
- [Background] Einhorn LH, Grunberg SM, Rapoport B, Rittenberg C, Feyer P. Antiemetic therapy for multiple-day chemotherapy and additional topics consisting of rescue antiemetics and high-dose chemotherapy with stem cell transplant: review and consensus statement. Support Care Cancer. 2011 Mar;19 Suppl 1:S1-4. doi: 10.1007/s00520-010-0920-z. Epub 2010 May 26. PMID 20505956
- [Background] Jordan K, Jahn F, Jahn P, Behlendorf T, Stein A, Ruessel J, Kegel T, Schmoll HJ. The NK-1 receptor-antagonist aprepitant in high-dose chemotherapy (high-dose melphalan and high-dose T-ICE: paclitaxel, ifosfamide, carboplatin, etoposide): efficacy and safety of a triple antiemetic combination. Bone Marrow Transplant. 2011 Jun;46(6):784-9. doi: 10.1038/bmt.2010.205. Epub 2010 Sep 13. PMID 20838387
- [Background] Pielichowski W, Barzal J, Gawronski K, Mlot B, Oborska S, Wasko-Grabowska A, Rzepecki P. A triple-drug combination to prevent nausea and vomiting following BEAM chemotherapy before autologous hematopoietic stem cell transplantation. Transplant Proc. 2011 Oct;43(8):3107-10. doi: 10.1016/j.transproceed.2011.08.010. PMID 21996238
- [Background] Stiff PJ, Fox-Geiman MP, Kiley K, Rychlik K, Parthasarathy M, Fletcher-Gonzalez D, Porter N, Go A, Smith SE, Rodriguez TE. Prevention of nausea and vomiting associated with stem cell transplant: results of a prospective, randomized trial of aprepitant used with highly emetogenic preparative regimens. Biol Blood Marrow Transplant. 2013 Jan;19(1):49-55.e1. doi: 10.1016/j.bbmt.2012.07.019. Epub 2012 Aug 1. PMID 22863840
- [Background] Khojainova N, Santiago-Palma J, Kornick C, Breitbart W, Gonzales GR. Olanzapine in the management of cancer pain. J Pain Symptom Manage. 2002 Apr;23(4):346-50. doi: 10.1016/s0885-3924(02)00378-0. PMID 11997204
- [Background] Bymaster FP, Falcone JF, Bauzon D, Kennedy JS, Schenck K, DeLapp NW, Cohen ML. Potent antagonism of 5-HT(3) and 5-HT(6) receptors by olanzapine. Eur J Pharmacol. 2001 Nov 2;430(2-3):341-9. doi: 10.1016/s0014-2999(01)01399-1. PMID 11711053
- [Background] Bloechl-Daum B, Deuson RR, Mavros P, Hansen M, Herrstedt J. Delayed nausea and vomiting continue to reduce patients' quality of life after highly and moderately emetogenic chemotherapy despite antiemetic treatment. J Clin Oncol. 2006 Sep 20;24(27):4472-8. doi: 10.1200/JCO.2006.05.6382. PMID 16983116
- [Background] Schmitt T, Goldschmidt H, Neben K, Freiberger A, Husing J, Gronkowski M, Thalheimer M, Pelzl le H, Mikus G, Burhenne J, Ho AD, Egerer G. Aprepitant, granisetron, and dexamethasone for prevention of chemotherapy-induced nausea and vomiting after high-dose melphalan in autologous transplantation for multiple myeloma: results of a randomized, placebo-controlled phase III trial. J Clin Oncol. 2014 Oct 20;32(30):3413-20. doi: 10.1200/JCO.2013.55.0095. Epub 2014 Sep 15. PMID 25225424
- [Background] Martin AR, Pearson JD, Cai B, Elmer M, Horgan K, Lindley C. Assessing the impact of chemotherapy-induced nausea and vomiting on patients' daily lives: a modified version of the Functional Living Index-Emesis (FLIE) with 5-day recall. Support Care Cancer. 2003 Aug;11(8):522-7. doi: 10.1007/s00520-003-0482-4. Epub 2003 Jun 25. PMID 12827483
- See also: Multinational Association Of Supportive Care In Cancer (MASCC)/European Society of Medical Oncology (ESMO) Antiemetic Guidelines 2013 — https://mascc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant: aprepitant plus standard anti-emetic regimen
  Aprepitant: Add aprepitant to anti-emetic regimen
- Olanzapine: olanzapine plus standard anti-emetic regimen
  Olanzapine: add olanzapine to anti-emetic regimen
Period: Overall Study
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine
Started | 18 | 25 | 9
Completed | 14 | 21 | 8
Not Completed | 4 | 4 | 1
Not completed — met exclusion criteria | 1 | 1 | 1
Not completed — Did not complete survey | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine | Total
Number analyzed (Participants) | 14 | 21 | 8 | 43
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58.5 [36 to 78] | 61 [30 to 72] | 54 [38 to 70] | 57.5 [30 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 11
  Male | 11 | 15 | 6 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 6 | 15 | 3 | 24
  African American | 5 | 5 | 4 | 14
  Hispanic | 2 | 0 | 0 | 2
  Asian | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 21 | 8 | 43
Conditioning Chemotherapy Regimen [Number; unit: participants]
  BEAM | 3 | 6 | 2 | 11
  1-day melphalan | 11 | 14 | 6 | 31
  2-day melphalan | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: no emesis and no rescue anti-emetic therapy
Time Frame: within 120 hours following melphalan administration; no emesis and no rescue therapy within 120 hours of melphalan administration (within 120 hours following last day of melphalan administration at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine
Number analyzed (Participants) | 14 | 21 | 8
Participants | 4 | 11 | 4

2. Secondary Outcome: Acute Complete Response
Description: no emesis or rescue therapy; Acute complete response defined as no emesis or rescue therapy required from time point of 0 to 24 hours following melphalan therapy administration
Time Frame: 0 (transplant time) to 24 hours post-transplant
Population: No data were collected or analyzed for this outcome.
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Delayed Complete Response
Description: no emesis or rescue therapy administered; Delayed complete response defined as no emesis or rescue therapy required from time point of 25 hours to 120 hours following melphalan therapy administration
Time Frame: 25-120 hours post-transplant
Population: No data were collected or analyzed for this outcome.
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for 3 years.
Arm/Group | Aprepitant | Olanzapine | Aprepitant Plus Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/14 | 21/21 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/14 | 3/21 | 1/8
Other Adverse Events (participants affected / at risk) | 0/14 | 0/21 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant (N=14) | Olanzapine (N=21) | Aprepitant Plus Olanzapine (N=8)
Mucositis (Gastrointestinal disorders) | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT02939287/Prot_SAP_ICF_003.pdf